CLINICAL TRIAL: NCT00916266
Title: Phase 1 Study of Autologous Bone Marrow Stem Cells Transplantation in Patients With Temporal Lobe Epilepsy
Brief Title: Autologous Bone Marrow Stem Cells Transplantation in Patients With Temporal Lobe Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto do Cerebro de Brasilia (Other)
Collaborators: Hospital Sao Lucas da PUCRS (Other); Instituto do Cerebro da PUCRS (Unknown)
Responsible Party: Principal Investigator, Jaderson Costa da Costa, MD, PhD, Hospital Sao Lucas da PUCRS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stem cells in Epilepsy
Record Dates: First submitted 2009-04-24; First posted 2009-06-09 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Epilepsy
Keywords: Seizure frequency; Hippocampal volume; Adverse effects
MeSH Terms: conditions — Epilepsy | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell transplantation (Experimental): Patients with refractory temporal lobe epilepsy that are transplanted with autologous bone marrow stem cells in order to provide seizure control.
  Interventions: Procedure: Stem cell transplantation

INTERVENTIONS:
Procedure: Stem cell transplantation — Transplantations with autologous bone marrow mononuclear stem cells by selective posterior cerebral artery angiography
  Other Names: BMMSC - Bone Marrow Mononuclear Stem Cells

SUMMARY:
This research investigates the use of autologous bone marrow stem cells for the treatment of medically refractory temporal lobe epilepsy patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate autologous bone marrow stem cells transplantation as a safe and potentially beneficial treatment for patients with temporal lobe refractory epilepsy. We are mainly evaluating seizure frequency, hippocampal volume an cognitive performance

ELIGIBILITY:
Inclusion Criteria:

* temporal lobe medically refractory epilepsy patients with hippocampal atrophy

Exclusion Criteria:

* under 18 or over 65 years old patients
* previous neurological surgery
* other neurodegenerative diseases

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
seizure frequency | 6 months

SECONDARY OUTCOMES:
adverse effects | 6 months
hippocampal volume | 6 months
cognitive performance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson C da Costa, MD, PhD, Principal Investigator — Instituto do Cerebro-PUCRS
Locations (1):
- Instituto do Cerebro, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Paglioli E, Palmini A, Portuguez M, Paglioli E, Azambuja N, da Costa JC, da Silva Filho HF, Martinez JV, Hoeffel JR. Seizure and memory outcome following temporal lobe surgery: selective compared with nonselective approaches for hippocampal sclerosis. J Neurosurg. 2006 Jan;104(1):70-8. doi: 10.3171/jns.2006.104.1.70. PMID 16509149
- [Background] Paglioli E, Palmini A, Paglioli E, da Costa JC, Portuguez M, Martinez JV, Calcagnotto ME, Hoefel JR, Raupp S, Barbosa-Coutinho L. Survival analysis of the surgical outcome of temporal lobe epilepsy due to hippocampal sclerosis. Epilepsia. 2004 Nov;45(11):1383-91. doi: 10.1111/j.0013-9580.2004.22204.x. PMID 15509239
- [Background] Friedrich MA, Martins MP, Araujo MD, Klamt C, Vedolin L, Garicochea B, Raupp EF, Sartori El Ammar J, Machado DC, Costa JC, Nogueira RG, Rosado-de-Castro PH, Mendez-Otero R, Freitas GR. Intra-arterial infusion of autologous bone marrow mononuclear cells in patients with moderate to severe middle cerebral artery acute ischemic stroke. Cell Transplant. 2012;21 Suppl 1:S13-21. doi: 10.3727/096368912x612512. PMID 22507676
- [Background] Costa-Ferro ZS, Vitola AS, Pedroso MF, Cunha FB, Xavier LL, Machado DC, Soares MB, Ribeiro-dos-Santos R, DaCosta JC. Prevention of seizures and reorganization of hippocampal functions by transplantation of bone marrow cells in the acute phase of experimental epilepsy. Seizure. 2010 Mar;19(2):84-92. doi: 10.1016/j.seizure.2009.12.003. Epub 2010 Jan 18. PMID 20080419
- [Background] Costa-Ferro ZS, Souza BS, Leal MM, Kaneto CM, Azevedo CM, da Silva IC, Soares MB, Ribeiro-dos-Santos R, Dacosta JC. Transplantation of bone marrow mononuclear cells decreases seizure incidence, mitigates neuronal loss and modulates pro-inflammatory cytokine production in epileptic rats. Neurobiol Dis. 2012 May;46(2):302-13. doi: 10.1016/j.nbd.2011.12.001. Epub 2011 Dec 11. PMID 22198377